CLINICAL TRIAL: NCT04361162
Title: Nivolumab and Ipilimumab and Radiation Therapy in Metastatic, Microsatellite Stable Pancreatic Cancer
Brief Title: Nivolumab + Ipilimumab + Radiation in MSS Pancreatic Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Theodore Sunki Hong, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-587
Record Dates: First submitted 2020-04-22; First posted 2020-04-24 (Actual); Last update posted 2022-09-08 (Actual); Status verified 2022-09

CONDITIONS: Pancreatic Cancer; Metastatic Pancreatic Cancer
Keywords: Pancreatic Cancer; Metastatic Pancreatic Cancer; Metastatic, Microsatellite Stable Pancreatic Cancer; Immunotherapy; Radiation therapy
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplasm Metastasis | interventions — Nivolumab; Ipilimumab; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Nivolumab + Ipilimumab + Radiation (Experimental): The research study procedures include screening for eligibility and study treatment including evaluations and follow up visits, (Study cycles are 6 weeks.)
  * Nivolumab via iv, at predetermined dose every 2 weeks for duration of study.
  * Ipilimumab via iv at a predetermined dose on day 1 of 4 study cycles.
  * Radiation treatments will be administered every other weekday or 2 days during week 1 of cycle 1.
  Interventions: Drug: Nivolumab; Drug: Ipilimumab; Radiation: Radiation

INTERVENTIONS:
Drug: Nivolumab — Nivolumab is a type of immunotherapy. Immunotherapy works by encouraging the body's own immune system to attack the cancer cells. Nivolumab work by stopping various molecules on cancer cells and body cells from working against the immune system's natural fight against cancer
  Other Names: Opdivo
Drug: Ipilimumab — Ipilimumab is a type of immunotherapy. Immunotherapy works by encouraging the body's own immune system to attack the cancer cells. Ipilimumab work by stopping various molecules on cancer cells and body cells from working against the immune system's natural fight against cancer
  Other Names: Yervoy
Radiation: Radiation — 3D Conformal Radiotherapy to shrink or kill tumors
  Other Names: RT

SUMMARY:
This research is being done to study the effects of the combination of ipilimumab, nivolumab, and radiation therapy in people with microsatellite stable pancreatic cancer.

The names of the study interventions involved in this study are:

* Ipilimumab
* Nivolumab
* Radiation Therapy

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial study testing the safety and effectiveness of the combination of ipilimumab, nivolumab, and radiation therapy.

The research study procedures include screening for eligibility, and study treatment including evaluations and follow up visits.

Participants will be in this research study for as long as the study interventions are safe and beneficial. Participants will then be followed for up to 5 years.

The names of the study interventions involved in this study are:

* Ipilimumab
* Nivolumab
* Radiation Therapy It is expected that about 30 people will take part in this research study.

Ipilimumab and Nivolumab are both antibodies. An antibody is a protein that attaches to other cells to fight off infection. The antibodies in ipilimumab work by not allowing cancer cell growth. The antibodies in nivolumab work by causing programmed cell death of the cancer cells. Radiation therapy may increase the likelihood of response to interventions like ipilimumab and nivolumab.

The U.S. Food and Drug Administration (FDA) has not approved ipilimumab and nivolumab for microsatellite stable pancreatic cancer. but they have been approved for other uses.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically or cytologically confirmed metastatic MSS adenocarcinoma of pancreatic origin
* Age >18 years.
* ECOG performance status <2
* Life expectancy of greater than 3 months
* Participants must have normal organ and marrow function as defined in Table 1, all screening labs should be performed within 14 days of protocol registration.
* Hematological

  * Absolute neutrophil count(ANC) ≥1000 /mcL
  * White blood count (WBC) ≥2000 /mcL
  * Platelets ≥75,000 / mcL
  * Hemoglobin ≥7.5 g/dL
* Renal

  * Serum creatinine: ≤ Serum creatinine ≤ 1.5 x ULN or creatinine clearance (CrCl) OR
  * Measured or calculated Creatinine clearance should be calculated per institutional standard: ≥ 40 mL/min (if using the Cockcroft-Gault formula below):
  * (GFR can also be used in place of creatinine or CrCl)

    * Female CrCl = (140 - age in years) x weight in kg x 0.85/ 72 x serum creatinine in mg/dL
    * Male CrCl = (140 - age in years) x weight in kg x 1.00/ 72 x serum creatinine in mg/dL
* Hepatic

  * Serum total bilirubin ≤ 1.5 X ULN (subjects with Gilbert Syndrome can have a total bilirubin <3 mg/dL
  * AST (SGOT) and ALT (SGPT) ≤ 3 X ULN OR ≤ 5 X ULN for subjects with liver metastases
* Coagulation

  * International Normalized Ratio (INR) or Prothrombin Time (PT) ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT is within therapeutic range of intended use of anticoagulants
  * Activated Partial Thromboplastin Time (aPTT) ≤2.5 X ULN unless subject is receiving anticoagulant therapy as long as PTT is within therapeutic range of intended use of anticoagulants
* Women of childbearing potential (WOCBP) must use appropriate method(s) of contraception. WOCBP should use an adequate method to avoid pregnancy for 5 months (30 days plus the time required for nivolumab to undergo five half-lives) after the last dose of investigational drug.
* Women of childbearing potential must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG)
* Women must not be breastfeeding
* Men who are sexually active with WOCBP must use any contraceptive method with a failure rate of less than 1% per year. Men receiving nivolumab and who are sexually active with WOCBP will be instructed to adhere to contraception for a period of 7 months after the last dose of investigational product. Women who are not of childbearing potential, ie, who are postmenopausal or surgically sterile as well as azoospermic men do not require contraception
* Ability to understand and the willingness to sign a written informed consent document.
* If applicable, stable dose of dexamethasone 1.5mg or prednisone <10mg for 7 days prior to initiation of treatment
* One previously unirradiated lesion amenable to radiotherapy 8 Gy x 3 and can meet dose constraints, and another unirradiated measurable lesion > 1 cm in size outside the radiation field that can be used as measurable disease. (Patients must have measurable tumor in addition to the one being radiated.)
* Patients must have progressed on at least 1 prior line of chemotherapy. Adjuvant or neoadjuvant therapy is permitted

Exclusion Criteria:

* Participants who have had chemotherapy, targeted small molecule therapy or study therapy within 14 days of protocol treatment, or those who have not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 2 weeks earlier. Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study. If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
* Participants who are receiving any other investigational agents.
* Patients are excluded if they have an active, known or suspected autoimmune disease other than those listed below. Subjects are permitted to enroll if they have vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger
* Patients are excluded if they have a condition requiring systemic treatment with either corticosteroids (dexamethasone 1.5mg or prednisone <10mg) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses dexamethasone 1.5mg or prednisone <10mg are permitted in the absence of active autoimmune disease. Subjects are permitted to use topical, ocular, intra-articular, intranasal, and inhalational corticosteroids (with minimal systemic absorption). Physiologic replacement doses of systemic corticosteroids are permitted, dexamethasone 1.5mg or prednisone <10mg. A brief course of corticosteroids for prophylaxis (eg, contrast dye allergy) or for treatment of non-autoimmune conditions (eg, delayed-type hypersensitivity reaction caused by contact allergen) is permitted.
* Patients are excluded if they have previously received anti-CTLA-4 therapy. Prior PD-1 or PDL1 therapy will be permitted.
* Has a known history of active TB (Bacillus Tuberculosis)
* Known HBV or HCV. (Patients are excluded if they are positive test for hepatitis B virus surface antigen (HBV sAg) or hepatitis C virus ribonucleic acid (HCV antibody) indicating acute or chronic infection).
* Patients are excluded if they have known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS).These participants are at increased risk of lethal infections when treated with marrow suppressive therapy. Appropriate studies will be undertaken in participants receiving combination antiretroviral therapy when indicated.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 5 months for woman and 7 months for men, after the last dose of trial treatment.
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin and squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
* Has known history of, or any evidence of active, non-infectious pneumonitis.
* Has an active infection requiring systemic therapy.
* Has received a live vaccine within 30 days of planned start of study therapy.Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.
* History of allergy to study drug components
* History of severe hypersensitivity reaction to any monoclonal antibody
* Uncontrolled brain metastases. Patients treated with radiation > 4 weeks prior with follow up imaging showing control are eligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-05-18 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | 6 weeks
  Overall response rate (ORR) will be evaluated by RECIST. Nivolumab and ipilimumab combined with radiation will be considered to have promising activity in metastatic MSS pancreatic cancer if at least 3 of 30 patients were to achieve CR or PR.

SECONDARY OUTCOMES:
Disease control rate (DCR) | Up to 5 yrs
  Disease control rate (DCR) will be based on RECIST and estimated with 95% confidence intervals based on the exact binomial distribution.
Number of Participants with Treatment Related Adverse Events as Assessed NCI CTCAE 5.0 guidelines | Up to 5 years
  Toxicity rates associated with the protocol treatment of nivolumab and ipilimumab combined with radiation will be summarized by category and grade.
Progression-free survival (PFS) | Up to 5 years
  Progression-free survival (PFS) is defined as the duration from the first day of protocol treatment to the earliest date of tumor progression by RECIST, appearance of new metastases, or death due to any cause. PFS time will be censored at the date of last follow-up for patients still alive with disease control. The PFS rate will be estimated using the Kaplan-Meier method with 95% confidence intervals based on the complementary log-log transformation.
Overall survival (OS) in patients | Up to 5 years
  Overall survival (OS) is defined as the duration from the first day of protocol treatment to the date of death due to any cause and will be censored at the date of last follow-up for patients still alive. The OS rate will be estimated using the Kaplan-Meier method with 95% confidence intervals based on the complementary log-log transformation.

CONTACTS AND LOCATIONS:
Overall Officials: Theodore S Hong, MD, Principal Investigator — Massachusetts General Hospital
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Partners Innovations team at http://www.partners.org/innovation